CLINICAL TRIAL: NCT02387879
Title: A Non-interventional, Multi-center, Observational Post Authorization Safety Study of Patients With Relapse/Refractory Multiple Myeloma Treated With Lenalidomide in Turkey
Brief Title: A Non-interventional,Observational Post Authorization Study of Patients With Multiple Myeloma Treated With Lenalidomide TR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-5013-PASS-TR
Record Dates: First submitted 2015-02-05; First posted 2015-03-13 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; PASS; Observational; Non-interventional; Relapse; Refractory; CC-5013; Lenalidomide; Turkey
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1: Subjects should be chosen among relapse/refractory multiple myeloma patients who have received at least one prior antimyeloma chemotherapy regimen (excluding treatment regimens with steroid only) with adequate dose and duration (≥2 cycles) or who have relapse/refractory multiple myeloma after stem cell transplantation.
  Patients who are eligible for the study will be consecutively enrolled in the study until the targeted patient number is reached. The responsible investigator will be requested to keep a log of subjects who are invited to enter the study. In the case of any of these subjects will not be enrolled in the study, this information will be documented together with its reason

SUMMARY:
CC-5013-PASS-TR/A non-interventional, multi-center, observational post authorization safety study of patients with relapsed/refractory multiple myeloma treated with Lenalidomide in Turkey.

The study is anticipated to last for approximately 8 years. Recruitment period will continue until 500 subjects have commenced the third cycle of treatment with lenalidomide.

DETAILED DESCRIPTION:
Objectives:

- Primary: To characterize and determine the incidence of adverse events of special interest; in subjects treated with Lenalidomide in real life setting in given indication.

- Secondary:

1. To observe the basic adverse event management approaches of physicians
2. To evaluate the effectiveness of Lenalidomide in given indication and to evaluate the prescription line.
3. To monitor the reasons of patients' noncompliance with lenalidomide usage recommended in Patient Information Leaflet.

Subjects will be recruited from approximately 36 hematology/oncology sites in Turkey. In all cases, the decision to treat the patient will be made prior to the decision to enter the subject into the study. All subjects enrolled will be prospectively followed up for up to 36 months, where feasible, following the end of observed treatment period. This 36 month observation period will start from end of treatment. The observation follow up period will end 36 months after the end of lenalidomide or background observed treatment period, or at time of death, withdrawal of consent, or loss to follow up. Following completion of treatment, subjects will be followed up after 30 days and then every 6 months to assess status.

Patients who are eligible and signed a consent form will be recruited consecutively. Subjects who temporarily discontinue treatment for any reason for more than 30 days will be withdrawn from treatment observation but will be observed for safety for up to 36 months (from the end of treatment). If the reason for discontinuation for subjects is due to an adverse event, the follow up of the adverse event will not be time limited and will continue until resolution or stabilization or when, in the opinion of the investigator, no additional useful information can be obtained from the event or the subject withdraws their consent to any more data being collected. Subjects will discontinue from the study if they switch to another treatment. No intervention will be performed to physician. Treatment will be according to physician's regular clinical practice.

All treatments will be prescribed by the treating investigator in accordance with regular clinical practice.

All assessments will be made according to the regular clinical practice of the treating investigator. Therefore if a parameter is requested on the case report form (CRF) but the investigator's normal practice is not to carry out such an assessment, then the field will not be completed.

Statistical Analysis:

Data from all subjects who receive at least one dose of treatment will be included in the safety analysis.

Adverse events will be classified using the MedDRA classification system. The severity of the toxicities will be graded according to the NCI CTCAE V. 4.03 whenever possible.

Adverse event frequency will be tabulated by body system and MedDRA term. In the by subject analysis, a subject having the same event more than once will be counted only once. Adverse events will be summarized by worst NCI CTCAE V. 4.03 grade.

Adverse events leading to death or to discontinuation from treatment, study-drug-related events, and serious adverse events will be listed separately.

The Kaplan-Meier procedures will be used to characterize time to onset and time to resolution for adverse events of special interest. Multivariate logistic regression will be used to determine the demographic and baseline characteristics most predictive of developing adverse events of interest. A forward selection stepwise procedure will be used to identify the subset of relevant factors.

Summary tables will also be provided for clinically relevant subgroups. Analyses will be undertaken to explore the course of neuropathy for subjects who have pre-existing neuropathy at baseline. Specifically, cross-tabulations will be used to summarize changes in severity observed during lenalidomide treatment and summary statistics will be provided for other relevant variables.

ELIGIBILITY:
Inclusion Criteria:

* Male or female multiple myeloma patients with ≥18 years of age.
* Subjects who understand and voluntarily sign an informed consent
* Subjects who are receiving lenalidomide treatment in combination with dexamethasone not longer than four weeks.

Exclusion Criteria:

* - Refusal to participate in the study.
* Patients who are currently on an interventional clinical trial
* Subjects who previously received lenalidomide treatment and whose treatment is ceased or who had a treatment interruption for four weeks or longer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It will continue until 500 subjects have commenced the third cycle of treatment with lenalidomide. As a condition of market authorization, subjects should be chosen among relapsed/refractory multiple myeloma patients who have received at least one prior antimyeloma chemotherapy regimen (excluding treatment regimens with steroid only) with adequate dose and duration (≥2 cycles) or who have relapsed/refractory multiple myeloma after stem cell transplantation. Patients who are eligible for the study will be consecutively enrolled in the study until the targeted patient number is reached. The responsible investigator will be requested to keep a log of subjects who are invited to enter the study. In the case of any of these subjects will not be enrolled in the study, this information will be documented together with its reason.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2013-12-25 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Up to 5 years
  Number of participants with Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Atiba-Davies, PhD, Study Director — Celgene
Locations (38):
- Turkey (Türkiye) (38):
  - Baskent University Adana Application and Research Hospital, Adana
  - Cukurova University Medical Faculty, Adana
  - Gulhane Military Medical Academy, Ankara
  - Ankara University Medical Faculty, Ankara
  - Ankara Numune Training and Research Hospital, Ankara
  - Diskapi Yildirim Beyazit Training and Research Hospital, Ankara
  - Dr. Abdurrahman Yurtaslan Ankara Onkology Training and Research Hospital, Ankara
  - Hacettepe University Medical Faculty, Ankara
  - Ankara Bayindir Hospital, Ankara
  - Baskent University Ankara Hospital, Ankara
  - Gazi University Medical Faculty, Ankara
  - Antalya Medstar Hospital, Antalya
  - Akdeniz University Medical Faculty, Antalya
  - Ali Osman Sonmez Oncology Hospital, Bursa
  - Uludag University Medical Faculty, Bursa
  - Pamukkale University Medical Faculty, Denizli
  - Dicle University Medical Faculty, Diyarbakır
  - Trakya University Medical Faculty, Edirne
  - Osmangazi University Medical Faculty, Eskişehir
  - Gaziantep University Medical Faculty, Gaziantep
  - Istanbul University Istanbul Medical Faculty, Istanbul
  - Istanbul University Cerrahpasa Medical Faculty, Istanbul
  - Bakırkoy Dr.Sadi Konuk Training and Research Hospital, Istanbul
  - Medipol University Medical Faculty, Istanbul
  - Kartal Training and Research Hospital, Istanbul
  - Marmara University Pendik Training and Research, Istanbul
  - Ege University Medical Faculty, Izmir
  - Dokuz Eylul University Medical Faculty, Izmir
  - Izmir Medical Park Hospital, Izmir
  - Erciyes University Medical Faculty, Kayseri
  - Kocaeli University Medical Faculty, Kocaeli
  - Necmettin Erbakan University Meram Medical Faculty, Konya
  - Inonu University Medical Faculty, Malatya
  - Celal Bayar University Medical Faculty, Manisa
  - Mersin University Medical Faculty, Mersin
  - Ondokuz Mayis University Medical Faculty, Samsun
  - Namik Kemal University Medical Faculty, Tekirdağ
  - Karadeniz Technical University Medical Faculty, Trabzon